CLINICAL TRIAL: NCT06876441
Title: A Randomized Controlled Trial to Evaluate the Effect of the Home-based Digital-assisted Dyadic Tai Chi (HDTC) Training Program on Cardiac Function Among Sedentary Individuals With Heart Failure (HF) and Care Burden of Their Caregivers.
Brief Title: Effect of the Home-based Digital-assisted Dyadic Tai Chi (HDTC) Training Program on Cardiac Function Among Sedentary Individuals With HF and Care Burden of Their Caregivers: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, XIE Yao Jie Grace, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20240904005
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure (HF)
Keywords: heart failure; Tai Chi; dyadic; cardiac function; care burden
MeSH Terms: conditions — Heart Failure; Caregiver Burden

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Participants (HF individuals and their caregivers) in this arm will receive a 30-min online comprehensive education and nurse-led support through telephone consultations in the aspects of symptom management, medication, dietary and exercise suggestions, psychosocial support, and regular monthly follow-up.
  Interventions: Other: Usual Care Group
- HDTC training program (Experimental): HF individual and caregiver dyads in the HDTC group will receive the usual care and also the HDTC training program, including a 30-minute educational seminar, a 1-hour dyadic coaching session, and 12-week Tai Chi training. The 24-form Yang-style Tai Chi will be adopted.
  Interventions: Behavioral: HDTC training program

INTERVENTIONS:
Behavioral: HDTC training program — Participants will receive usual care plus HDTC training program, including four parts: (1)30-minute educational seminar via WeChat: provide disease knowledge, propose strategies to replace sedentary behavior, and introduce Tai Chi. (2)1-hour online nurse-lead dyadic coaching session: introduce dyadic Tai Chi, clarify the roles and responsibilities, and establish a shared goal among dyads. (3)1-hour preliminary Tai Chi training session: face-to-face, introduce online Tai Chi learning, demonstrations on using heart rate monitor. (4)12-week Tai Chi training: Dyads learn Tai Chi following Tai Chi master online. The frequency gradually increased from 2 to 3 classes per week and duration extending from 30 to 50 minutes. Subsequently, they will practice Tai Chi with the master once a week and follow instructional videos twice a week, with each session lasting 50 minutes. The finalized contents will be determined based on the pilot RCT.
  Arms: HDTC training program
Other: Usual Care Group — HF-caregiver dyads in the control group will receive the usual care, including a 30-min online comprehensive education and nurse-led support through telephone consultations in the aspects of symptom management, medication, dietary and exercise suggestions, psychosocial support, and regular monthly follow-up every month.
  Arms: Usual care

SUMMARY:
Firstly, we will conduct a pilot RCT before this full scale RCT to assess the feasibility, acceptability, and preliminary efficacy of the HDTC training program. If the HDTC training program is feasible and acceptable, this full scale will then conducted based on the refined protocol. The full scale RCT aims to assess the effectiveness of the HDTC training program in improving cardiac function and secondary outcomes among sedentary heart failure individuals, while simultaneously reducing care burden and improving other outcomes for their caregivers.

DETAILED DESCRIPTION:
The pilot part is a two-arm parallel, single-blinded randomized controlled trial. 20 HF dyads will be enrolled and attend the 12 weeks intervention. The full scale RCT is a two-arm parallel, single-blinded randomized controlled trial. A total of 118 HF individuals and 118 caregivers will be enrolled and allocated to the HDTC group and the control group in a 1:1 ratio. Participants in the control group will receive usual care. Those in the HDTC group will attend usual care plus the HDTC training program, including a 30-minute educational seminar, a 1-hour dyadic coaching session, and 12-week Tai Chi training. Data on cardiac function, exercise tolerance, exercise self-efficacy, fear of activity, sedentary behavior, hospital admission, health-related quality of life, depression, anxiety, stress, and mutuality for HF individuals, as well as care burden, quality of life, depression, anxiety, stress, and mutuality of caregivers, will be collected at baseline (T0), 4 weeks (T1) and 12 weeks (T2) after the intervention. The intention-to-treat analysis (ITT), modified ITT analysis, and per-protocol analysis will be conducted. The generalized estimating equation (GEE) model will be used to measure changes in outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* HF individuals:

  * aged 18 to 75 years
  * diagnosed with CHF based on the Chinese Guidelines for Diagnosis and Treatment of Heart Failure 2024
  * categorized as NYHA class I, II or III
  * 6MWD >150 meters (mild to moderate HF)
  * stable phase of disease in the past four weeks and capable of independently practice Tai Chi without any musculoskeletal disorders that may impede joint movement
  * sit more than 8 h/d in the past month
  * own a smartphone
  * volunteer to participate and provide informed consent.
* caregivers:

  * age ≥18 years old
  * primary caregiver at home, who has emotional ties or social obligations with HF individuals and provides daily care
  * able to exercise Tai Chi without help
  * volunteer to participate and provide informed consent.

Exclusion Criteria:

* HF individuals:

  * plan to undergo surgery within the next 6 months
  * have severe comorbidities, such as cancer, liver or kidney failure, or diagnosed psychiatric disorders
  * plan to be admitted to a nursing home or other care facilities
  * regularly practice Tai Chi or engaging in other forms of exercise in the past 3 months (at least 3 times per week, at least 20 minutes of regular exercise each time)
  * currently participate in similar or related studies.
* caregivers: · formal caregivers, such as nurses, will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
cardiac function of HF individuals | From enrollment to the end of intervention at 4 weeks and 12 weeks
  The primary outcome of this study is the cardiac function, measured by LVEF. LVEF is a crucial parameter for assessing cardiac function. It is an echocardiographic measure that reflects cardiac function by indicating the percentage of blood ejected from the left ventricle with each heartbeat. Three-dimensional echocardiography will be employed to measure LVEF.
  For the pilot RCT, the primary outcome is the feasibilty and acceptability measuring by recruitment period, recruitment rate, attendance rate and adherence rate of online Tai Chi classes, attrition rate, and dyads opinions about the intervention based on the Theoretical Framework of Acceptability.

SECONDARY OUTCOMES:
exercise tolerance of HF individuals | From enrollment to the end of intervention at 4 and 12 weeks
  The 6MWT will be used to assess exercise tolerance.
sedentary behavior of HF individuals | From enrollment to the end of intervention at 4 and 12 weeks
  HF individuals' sedentary behavior will be assessed using the International Physical Activity Questionnaire-Short Form (IPAQ-SF).
hospital admission of HF individuals | From enrollment to the end of intervention at 12 weeks
  The HF individual's hospital admission status will be presented based on the number of hospital admissions during the intervention period, including emergency visits.
Health-related QoL of HF individuals | From enrollment to the end of intervention at 4 and12 weeks
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a specific and commonly used scale for measuring QoL among HF patients, which will be used to assess QoL.
care burden of caregivers | From enrollment to the end of intervention at 4 and 12 weeks
  The Chinese version of the Zarit Caregiver Burden Interview (ZBI), will be used to measure caregivers' perceived burden of providing care.
QoL of caregivers | From enrollment to the end of intervention at 4 and 12 weeks
  The Family Caregiver Quality of Life (FAMQOL) is a specific instrument designed by Nauser in 2011 to assess the QoL among caregivers of HF patients.

OTHER OUTCOMES:
Exercise self-efficacy of HF individuals | From enrollment to the end of intervention at 4 and 12 weeks
  Exercise self-efficacy will be assessed utilizing the Self-Efficacy for Exercise Scale (SEE) , which specifically measures an individual's confidence in performing exercise despite various barriers. The scale consists of 9 items with scores ranging from 0 to 90, with higher score indicating greater confidence in participating in exercise activities.
Fear of Activity of HF individuals | From enrollment to the end of intervention at 4 and 12 weeks
  Fear of Activity in Patients with Chronic Heart Failure (Fact-CHF) will be used to assess HF patients' fear of exercise. This scale consists of 15 items, using a 5-point Likert scale where 0 represents 'never' and 4 represents 'always'. The total score ranges from 0 to 60, with higher scores indicating higher levels of fear.
mutuality of HF-caregiver dyads | From enrollment to the end of intervention at 4 and 12 weeks
  Mutuality, is a dyadic-level variable influencing caregiver's contribution to HF self-care, with a good relationship improving the dyadic health of both patients and caregivers. The Mutuality Scale (MS) will be used, containing 15 items categorized into four dimensions: love and affection, shared values, shared enjoyable activities, and reciprocity. Responses are rated using a 5-point Likert type (0=not at all, 4=quite a lot). The mean item score will be computed as the final score, ranging from 0 to 4, with a higher score denoting better mutuality.
depression, anxiety, and stress of HF-caregiver dyads | From enrollment to the end of intervention at 4 and 12 weeks
  The Depression Anxiety Stress Scales-21 (DASS-21) will be used to assess the severity of psychological distress about depression, anxiety, and stress over the preceding week of both HF patients and their caregivers. Each of the three DASS-21 subscales contains 7 items, with a total of 21 items. A Likert scale ranging from 0 to 3 is employed, with recommended cut-off scores of 9, 7, and 14 for depression, anxiety, and stress, respectively. The higher the score, the higher the level of anxiety, depression, and stress.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No